CLINICAL TRIAL: NCT05672966
Title: A Phase I, First-in-human, Randomized, Observer-blinded, Placebo-controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of BV601 in Healthy Adult Volunteers
Brief Title: Phase I Clinical Trial of a Candidate HPV Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan BravoVax Co., Ltd. (Industry)
Collaborators: Shanghai BravoBio Co., Ltd. (Unknown); Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BV-C601-202201
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV Vaccine; Phase I; BV601
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1-BV601DP(Low dose HPV vaccine with adjuvant) (Experimental): Subjects received low dose of BV601DP
  Interventions: Biological: Human papillomavirus (HPV) Vaccine
- 1-BV601DPP(Low dose HPV vaccine without adjuvant) (Experimental): Subjects received low dose of BV601DPP
  Interventions: Biological: Human papillomavirus (HPV) Vaccine
- 1-Placebo (Placebo Comparator): Subjects received placebo
  Interventions: Biological: Placebo
- 2-BV601DP(High dose HPV vaccine with adjuvant) (Experimental): Subjects received high dose of BV601DP
  Interventions: Biological: Human papillomavirus (HPV) Vaccine
- 2-BV601DPP(High dose HPV vaccine without adjuvant) (Experimental): Subjects received high dose of BV601DPP
  Interventions: Biological: Human papillomavirus (HPV) Vaccine
- 2-Placebo (Placebo Comparator): Subjects received placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Human papillomavirus (HPV) Vaccine — 0.5mL, Intramuscular
  Other Names: BV601
  Arms: 1-BV601DP(Low dose HPV vaccine with adjuvant); 1-BV601DPP(Low dose HPV vaccine without adjuvant); 2-BV601DP(High dose HPV vaccine with adjuvant); 2-BV601DPP(High dose HPV vaccine without adjuvant)
Biological: Placebo — 0.5mL, Intramuscular
  Arms: 1-Placebo; 2-Placebo

SUMMARY:
This is a Phase I, first-in-human, randomized, observer-blinded, placebo-controlled, dose escalation study to evaluate the safety, tolerability, and immunogenicity of BV601 (a HPV Vaccine) in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years (inclusive) at the time of Screening Visit.
* In good general health, with no significant medical history, and have no clinically significant abnormalities on vital signs, physical examination, laboratory tests, and ECG at Screening Visit and before the first vaccination of IP at the discretion of the Investigator(s) or designee.
* Body Mass Index (BMI) of ≥ 18.0 and ≤ 32.0 (BMI will be calculated by weight in kilograms [kg]/square of height in meters [m2]) and weigh at least 50 kg at Screening Visit.
* Able and willing to comply with all study requirements and study procedures.
* Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.
* Male and female of childbearing age should agree to take effective contraception measures

Exclusion Criteria:

* Physical or psychological medical histories (within 3 months prior to Screening Visit) or ongoing conditions of any clinically significant hepatic (eg, active liver disease, hepatic impairment), renal/genitourinary (eg, renal impairment), gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological, hematological disease, and/or any other medical conditions which, at the discretion of the Investigator(s), may jeopardize the safety of the participants and/or effect the results of the study.
* Histories or on-going conditions of immune function impaired, congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases.
* Histories or on-going conditions of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago.
* History of abnormal cervical biopsy results (showing cervical intraepithelial neoplasia or worse) or cervical disease (ie, surgical treatment for cervical lesions) within 5 years prior to Screening Visit.
* History of a positive test for HPV infection.
* Histories of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents.
* Loss of spleen or functional spleen, and/or removal of spleen caused by any situation
* Body temperature before vaccination ≥ 38℃ for ear or temporal artery temperature or ≥ 37.2 ℃ for armpit temperature before vaccination.
* Systolic blood pressure ≥ 140 mmHg and/or a diastolic blood pressure ≥ 90 mmHg before vaccination.
* Receipt of systemic immunosuppressants or immune-modifying drugs for > 14 days in total within 6 months prior to Screening Visit (for corticosteroids ≥ 20 mg/day of prednisone equivalent). Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Receipt of immunoglobulins and/or any blood products within the 3 months prior to the first vaccination or planned administration during the study period.
* Receipt of any HPV vaccination within 3 months prior to the first vaccination. Receipt of any vaccination other than HPV vaccination within 30 days prior to first vaccination. Plan to receive any vaccination within 7 days prior to the secondary or third IP vaccination. Plan to receive any vaccination within 30 days after the first, secondary, or third IP vaccination.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first vaccination of IP.
* Use of (or anticipated use of) any prescription drugs (other than hormonal contraception; oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones, a vaginal ring, or an IUD), over the counter (OTC) medication, or herbal remedies 2 weeks prior to dosing and during course of study, unless the medication will not affect the safety and efficacy evaluations in the study at the discretion of the Investigator(s).
* Regular alcohol consumption defined as > 21 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit or a 125 mL glass of wine).
* Positive toxicology panel (urine test including qualitative identification of barbiturates, THC, amphetamines, benzodiazepines, opiates, and cocaine).
* Positive results of hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), HIV antibody, HPV, SARS-CoV-2, and pregnancy test.
* Pregnancy or breast feeding or plan to get pregnant or breastfeed during the study.
* Anything that the Investigator(s) considers that may jeopardise the safety of the participant, prevent complete participation in the study, or compromise interpretation of study data.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety in terms of solicited adverse events | within 7 days after each vaccination
  Occurrence of solicited AEs of each subject
Safety in terms of solicited systemic AEs | within 7 days after the first vaccination
  Occurrence of solicited systemic AEs of each subject
Safety in terms of dose-limiting toxicity (DLT) | within 30 days after the first vaccination
  Percentage of participants with dose-limiting toxicity
Safety in terms of unsolicited AEs | 365 days after the first vaccination
  Percentage of participants with unsolicited AEs
Safety in terms of all solicited and unsolicited AEs | 365 days after the first vaccination
  Frequency and severity of solicited and unsolicited AEs

SECONDARY OUTCOMES:
Immunogencity in terms of GMT by ELISA | Days 1, 31, 61, 91, 121, 181, 211, and 365
  GMT of anti-L2 immunoglobulin G (IgG) antibody responses
Immunogencity in terms of Nab | Days 1, 31, 61, 91, 121, 181, 211, and 365
  GMT of anti-HPV 6, 11, 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68, and 73 type specific serum neutralizing antibody (NAb) response
Immunogencity in terms of Seroconversion rate | Days 1, 31, 61, 91, 121, 181, 211, and 365
  Seroconversion rate of anti-L2 IgG antibody and anti-HPV 6, 11, 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68, and 73 type-specific serum Nab

CONTACTS AND LOCATIONS:
Locations (1):
- Paratus Clinical Research Canberra, Canberra, Australia

REFERENCES:
- [Derived] Han Z, Wang S, Mu T, Zhao P, Song L, Zhang Y, Zhao J, Yin W, Wu Y, Wang H, Gong B, Ji M, Roden RBS, Yang Y, Klein M, Wu K. Vaccination with a Human Papillomavirus L2 Multimer Provides Broad Protection against 17 Human Papillomavirus Types in the Mouse Cervicovaginal Challenge Model. Vaccines (Basel). 2024 Jun 20;12(6):689. doi: 10.3390/vaccines12060689. PMID 38932417